CLINICAL TRIAL: NCT06576479
Title: Validation of the Therapeutic Effect and Safety of a Specialized Oral Supplement on the Nutritional Status and Quality of Life in Patients with Chronic Kidney Disease Without Replacement Therapy: (Grade G3a, G3b, G4 and G5)
Brief Title: Effect of a Specialized Oral Supplement on Nutritional Status and Quality of Life in Non-dialysis CKD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NIN Institute (Industry)
Collaborators: Hospital Civil de Guadalajara (Other)
Responsible Party: Principal Investigator, Ari Cisneros-Hernández, Investigador Principal, Hospital Civil de Guadalajara
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: NI0001/24
Record Dates: First submitted 2024-08-19; First posted 2024-08-28 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Chronic Kidney Diseases; Protein-Energy Malnutrition
Keywords: chronic kidney disease; PEW; nutrition
MeSH Terms: conditions — Renal Insufficiency, Chronic; Protein-Energy Malnutrition | interventions — Nutrition Assessment

STUDY DESIGN:
Intervention Model Description: The intervention group receives specialized oral nutritional supplements plus nutritional counseling, the control group only receives nutrition counseling. Both groups receive laboratory studies (blood and urine) as well as body composition analysis with the use of electronic bioimpedance.
Who Masked: Investigator
Masking Description: The participant takes a random envelope without seeing, which the researcher receives and is automatically assigned the group in which he will remain until satisfactorily finished.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm Intervention (Experimental): Intervention group: The specialized oral supplement is provided, with the consumption of 1 serving (70g-dissolved in 237 ml natural water) per day in conjunction with individualized nutritional counseling. For 4 months
  Interventions: Dietary Supplement: Nutritious Shake
- Arm no Intervention (Other): Control group: They receive specialized nutrition considering the recommendations of the clinical practice guidelines for CKD. For 4 months
  Interventions: Behavioral: Nutritional counseling

INTERVENTIONS:
Dietary Supplement: Nutritious Shake — Powder 70 g/d diluted in 237 ml natural water
  Other Names: NIN
  Arms: Arm Intervention
Behavioral: Nutritional counseling — Specialized nutritional recommendations for CKD
  Arms: Arm no Intervention

SUMMARY:
Patients whit chronic kidney disease (CKD) there is a high prevalence of nutritional disorders and negative changes in body composition, which is strongly associated with an increased risk of morbidity and mortality.

DETAILED DESCRIPTION:
Epidemiological studies have reported that between 30 and 50% of patients with kidney disease show signs of malnutrition and that specifically in patient with CKD in stages 4-5 without replacement therapy, the prevalence of protein energy wasting (PEW) can be up to 45%.

Many factors influence the development of PEW, however, one main factor is insufficient intake of energy and macronutrients. The main obstacle that prevents the patient from meeting their nutritional requirements is the presence of gastrointestinal symptoms. In addition to this, dietary restrictions, lack of adherence to eating plans and the presence of digestive and psychological abnormalities of the patient, contribute directly to the patient directly contribute to insufficient energy and protein intake. Therefore, there is a need for evidence-based nutritional treatment strategies that facilitate the patient's achievement of their nutritional requirements and maintain or improve their nutritional supplements in patients with CKD has been shown to be a good treatment strategy.

Specifically in patients with CKD without replacement therapy, it has been observed that the use of specialized nutritional supplements can contribute to increasing their energy, fat, and fiber intake, while at the same time achieving a decrease in protein intake without causing any change in serum minerals or electrolytes.

This project will provide practical information for the validation of the therapeutic effect of a new specialized food supplement on the nutritional status and quality of life in patients with CKD without replacement therapy, which will be useful both for health professionals and for the patients themselves.

MAIN OBJETIVE:

To assess the effect and safety of the use of a specialized food supplement on the nutritional status and quality of life of patients with CKD and PEW without replacement therapy.

STUDIO DESING:

Randomized, blinded clinical trial with an intervention period of 4 months.

PROCESS:

1. Identify those patients who are candidates to participate in the clinical trial.
2. Review the inclusion and exclusion criteria.
3. Invite identified patients to participate in the clinical trial.

Pre - Nutritional wash out appointment - nutritionist

1. Evaluate inclusion criteria.
2. Review and sign the informed consent.
3. Perform evaluation to indicate a personalized meal plan.
4. Deliver a meal plan.
5. Schedule in 30 days for your next nutritional appointment.

0 - Full Assessment Nutritional Appointment - Nutritionist

1. Evaluate adherence to the meal plan (percentage of adequacy of energy and protein consumption from 70% to 130%).
2. Assign an intervention group randomly (sealed envelope).
3. Perform an evaluation of nutritional status, quality of life and body composition.

   Offer nutritional treatment according to the assigned intervention group.
4. Schedule an immediate appointment for laboratory tests of blood and urine.
5. Schedule in 30 days for your next nutritional appointment.

month 1 - Nutritional monitoring appointment - nutritionist

1. Evaluate adherence to the eating plan.
2. Offer nutritional treatment according to the assigned intervention group.
3. Schedule in 30 days for your next nutritional appointment.
4. Make an appointment a few days before your next nutritional appointment to perform blood and urine lab tests.

month 2 - Full Assessment Nutritional Appointment - Nutritionist

1. Perform an evaluation of nutritional status, quality of life and body composition.
2. Offer nutritional treatment according to the assigned intervention group.
3. Schedule in 30 days for your next nutritional appointment.

month 3 - Nutritional monitoring appointment - nutritionist

1. Evaluate adherence to the eating plan.
2. Offer nutritional treatment according to the assigned intervention group.
3. Schedule in 30 days for your next nutritional appointment. 4.3 - Nutritional monitoring appointment - nutritionist

5.Evaluate adherence to the eating plan. 6.Offer nutritional treatment according to the assigned intervention group. 7.Schedule in 30 days for your next nutritional appointment. 7.1Schedule a few days before your nutritional appointment for blood and urine lab tests.

month 4 - Full Assessment Nutritional Appointment - Nutritionist

1. Perform an evaluation of nutritional status, quality of life and body composition.
2. Offer nutritional treatment according to the assigned intervention group.

SAMPLE SIZE: 50 participants

STATISTIC ANALYSIS:

For the comparison of proportions between the groups, it will be done with X2 or Fisher's exact test and to compare quantitative variables, Student's T or Mann-Whitney U will be used. For the intra-group comparisons, Mc Nemar will be used for the qualitative variables and Anova for repeated samples or Friedman's Anova for the quantitative variables. For the analysis of the interaction or intervening variables, a stratified statistical analysis will be carried out, using contingency tables and the Mantel-Haenszel method. The results will be considered statistically significant if the value of p <0.05.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age
* Patients with diabetic kidney with eGFR <60 ml / min / 1.73m2 and ≥15 ml / min / 1.73m2, (stage G3a, G3b and G4 respectively)
* Patients with protein energy expenditure (defined by serum albumin < 3.8 g/dl)
* Patients with protein energy expenditure (defined by 24-hour recall less than a dietary protein intake <0.6 g/kg/d or have a consumption <25 kcal/kg/d
* Patients who can read and write (or primary caregiver)
* Domicile within the metropolitan area

Exclusion Criteria:

* Previous hospitalizations in the last month
* Patients with serious complications (chronic infection, septicemia, cancer, HIV, Alzheimer's, uncontrolled heart failure, liver failure, cerebrovascular syndrome, malabsorption syndrome, or allergy to any ingredient in the nutritional supplement)
* Patients with actual consumption of food supplements and / or keto analogues.

Elimination Criteria:

* Failure to attend nutritional assessment and biochemical testing at baseline, 2 months, and end of the study.
* Failure to take the supplement >10% (>12 failed doses).
* Diagnosis of any comorbidity during the intervention period.
* Initiation of replacement therapy.
* Identification of adverse effects.
* Withdrawal of voluntary participation by the patient.
* Death.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-07-10 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Serum Albumin (g/dl) | baseline intervention and 4 months
  Changes in serum albumin (g/dl) for all the patients at baseline and month 4.
Dietary intake (kcal/kg/day) | baseline intervention and 4 months
  Changes in dietary caloric intake of patients at baseline and month 4.

SECONDARY OUTCOMES:
Adherence to nutritional treatment | baseline intervention and 4 months
  Number of patients who manage to adhere correctly to the treatment, applying a Likert scale.
Adverse effects | baseline intervention and 4 months
  Number of patients who present adverse effects during the intervention, considering frequency and intensity by applying SAS (symptom assessment scale) and Bristol Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Paola Azucena Alvarado Pelayo, Bachelor, Principal Investigator — Hospital Civil Fray Antonio Alcalde
Locations (1):
- Hospital Civil Fray Antonio Alcalde, Guadalajara, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Carrero JJ, Stenvinkel P, Cuppari L, Ikizler TA, Kalantar-Zadeh K, Kaysen G, Mitch WE, Price SR, Wanner C, Wang AY, ter Wee P, Franch HA. Etiology of the protein-energy wasting syndrome in chronic kidney disease: a consensus statement from the International Society of Renal Nutrition and Metabolism (ISRNM). J Ren Nutr. 2013 Mar;23(2):77-90. doi: 10.1053/j.jrn.2013.01.001. PMID 23428357
- [Background] Riella MC. Nutritional evaluation of patients receiving dialysis for the management of protein-energy wasting: what is old and what is new? J Ren Nutr. 2013 May;23(3):195-8. doi: 10.1053/j.jrn.2013.01.023. PMID 23611546
- [Background] Perez-Torres A, Gonzalez Garcia ME, San Jose-Valiente B, Bajo Rubio MA, Celadilla Diez O, Lopez-Sobaler AM, Selgas R. Protein-energy wasting syndrome in advanced chronic kidney disease: prevalence and specific clinical characteristics. Nefrologia (Engl Ed). 2018 Mar-Apr;38(2):141-151. doi: 10.1016/j.nefro.2017.06.004. Epub 2017 Jul 26. English, Spanish. PMID 28755901
- [Background] Kovesdy CP, Kopple JD, Kalantar-Zadeh K. Management of protein-energy wasting in non-dialysis-dependent chronic kidney disease: reconciling low protein intake with nutritional therapy. Am J Clin Nutr. 2013 Jun;97(6):1163-77. doi: 10.3945/ajcn.112.036418. Epub 2013 May 1. PMID 23636234
- [Background] Zhang X, Bansal N, Go AS, Hsu CY. Gastrointestinal symptoms, inflammation and hypoalbuminemia in chronic kidney disease patients: a cross-sectional study. BMC Nephrol. 2015 Dec 11;16:211. doi: 10.1186/s12882-015-0209-z. PMID 26651991
- [Background] Paes-Barreto JG, Silva MI, Qureshi AR, Bregman R, Cervante VF, Carrero JJ, Avesani CM. Can renal nutrition education improve adherence to a low-protein diet in patients with stages 3 to 5 chronic kidney disease? J Ren Nutr. 2013 May;23(3):164-71. doi: 10.1053/j.jrn.2012.10.004. Epub 2012 Nov 27. PMID 23194841
- [Background] Tomayko EJ, Kistler BM, Fitschen PJ, Wilund KR. Intradialytic protein supplementation reduces inflammation and improves physical function in maintenance hemodialysis patients. J Ren Nutr. 2015 May;25(3):276-83. doi: 10.1053/j.jrn.2014.10.005. Epub 2014 Nov 25. PMID 25455421
- [Background] Kalantar-Zadeh K, Cano NJ, Budde K, Chazot C, Kovesdy CP, Mak RH, Mehrotra R, Raj DS, Sehgal AR, Stenvinkel P, Ikizler TA. Diets and enteral supplements for improving outcomes in chronic kidney disease. Nat Rev Nephrol. 2011 May 31;7(7):369-84. doi: 10.1038/nrneph.2011.60. PMID 21629229
- [Background] Cheu C, Pearson J, Dahlerus C, Lantz B, Chowdhury T, Sauer PF, Farrell RE, Port FK, Ramirez SP. Association between oral nutritional supplementation and clinical outcomes among patients with ESRD. Clin J Am Soc Nephrol. 2013 Jan;8(1):100-7. doi: 10.2215/CJN.13091211. Epub 2012 Oct 18. PMID 23085729
- [Background] Satirapoj B, Prapakorn J, Punpanich D, Pongsuparbchon C, Supasyndh O. The effect of ONCE Renal on minerals and electrolytes in predialysis patients with chronic kidney disease. Int J Nephrol Renovasc Dis. 2016 Apr 5;9:81-6. doi: 10.2147/IJNRD.S98179. eCollection 2016. PMID 27103839